CLINICAL TRIAL: NCT03417128
Title: Nutrition and Lifestyle Behaviours in Cardiometabolic Syndrome: Development of a Community-specific Peer-support Programme.
Brief Title: Nutrition and Lifestyle Behaviour Peer Support Program Among Malaysian Adults With Metabolic Syndrome (PERSUADE)
Acronym: PERSUADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Amutha Ramadas, Dr, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CF16/56 - 2016000022
Record Dates: First submitted 2017-12-26; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Metabolic Syndrome X; Nutritional and Metabolic Diseases; Health Behavior
MeSH Terms: conditions — Metabolic Syndrome; Nutritional and Metabolic Diseases; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group will receive a one-time personalised nutrition and lifestyle advised based from the Malaysian Dietary Guideline 2010. They will be assured to be followed up twice for the next six month.
- Peer support (Experimental): This group will receive a continuous three-months, peer-led nutrition and lifestyle behaviour intervention through a series of peer gathering.
  Interventions: Behavioral: Peer support

INTERVENTIONS:
Behavioral: Peer support — Participants residing in the location selected to be intervene will to form at minimum 4 peer groups. This group will receive a continuous three-months, peer-led nutrition and lifestyle behaviour intervention through a series of peer gathering. Two participants from each peer group will be selected as the peer leader (PL). PL will be trained to deliver the content of PERSUADE modules and will be responsible to run a weekly peer gathering with their respective groups for the following three months.
  Arms: Peer support

SUMMARY:
The outlook of a community-based intervention targeting nutrition and lifestyle behaviour modification among adults with metabolic syndrome (MetS) has not been fully explored. The primary aim of this study (PERSUADE) is to evaluate the effect of the peer support intervention on the clinical outcomes MetS components followed by improvements in the participants' dietary practices, physical activity levels and lifestyle behaviours. The program constructed using information obtained from the published clinical and dietary guideline in Malaysia.

DETAILED DESCRIPTION:
Aim: To develop and assess a three-month, group-based community peer support program for Malaysian adults with MetS.

Method:

The PERSUADE module will be constructed using the Health Belief Model (HBM) to address relevant health messages from the appropriate guidelines and recent literature evidence on MetS among Malaysian adults. Following that, a minimum sample of 96 Malaysian adults with MetS will be randomised, either to the control group, who will receive one-time standard nutrition and lifestyle advice or the intervention group, who will participate in a three-month peer support program using the PERSUADE module. The participants will be followed up for three months post-intervention with data collection scheduled at baseline, 3-month and 6-month.

PERSUADE is thoroughly designed using the current available guidelines informed with gathered inputs on motivations and barriers towards healthy lifestyle among Malaysians. The program aims to improve the clinical outcomes of MetS component among participants of the intervention group, besides the impact of the peer support intervention on the dietary practices, physical activity levels and lifestyle behaviours of those participants. The successful outcome of this study can be an initiator for policy makers to encourage more rigorous promotion of such community-based programmes in the country.

ELIGIBILITY:
Inclusion Criteria:

1. Physically healthy men and women who are ≥ 18 years old.
2. Literate with a fair command of Bahasa Melayu and/or English.
3. Metabolic syndrome status confirmed according to Harmonised Criteria.
4. Willing to attend weekly peer gathering sessions.

Exclusion Criteria:

1. Pregnant, lactating or intend to become pregnant during the study period.
2. Diagnosed with Type 1 Diabetes Mellitus (T1DM)
3. Any predisposing condition compromising the quality of life or ability to participate according to protocol.
4. Reported severe complications (chronic heart disease, cerebrovascular disease, diagnosed HIV/AIDS, cancer, emphysema, chronic liver or kidney disease) that would affect the participants' ability to follow the participation in peer activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-03-15 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline waist circumference at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  Waist circumference will be measured in centimeters using a body tape.
Changes from baseline systolic blood pressure at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  Systolicblood pressure will be expressed in mmHg using an automated blood pressure monitor (OMRON, Japan).
Changes from baseline diastolic blood pressure at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  Diastolic blood pressure be expressed in mmHg using an automated blood pressure monitor (OMRON, Japan).
Changes from baseline fasting blood triglyceride levels at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  Fasting blood triglyceride levels will be measured in mmol/l using a blood lipid meter (Cardiocheck PA, USA).
Changes from baseline fasting blood HDL-cholesterol levels at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  Fasting blood HDL-cholesterol levels will be measured in mmol/l using a blood lipid meter (Cardiocheck PA, USA).
Changes from baseline fasting blood sugar levels at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  Fasting blood glucose levels will be measured in mmol/l using a glucometer (B.Braun, Germany).

SECONDARY OUTCOMES:
Changes from baseline dietary intake at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  A 3-days 24 hour dietary recall will be done and analysed using a software (Nutritionist Pro, Axxya System, USA). Total calories intake (kcal) and macronutrients profile; carbohydrate, fat and protein (grams and percentage of daily energy intake) will be sought.
Changes from baseline physical activity levels at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  Physical activity levels will be measured using a validated short form International Physical Activity Questionnaire (IPAQ) and will be expressed in metabolic equivalent quotient (METS).
Changes from baseline lifestyle behaviour at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  A short questionnaire will be developed to gather information of sleep duration, smoking and alcohol consumption.
Changes from baseline health-related quality of life at post-intervention and 3 months follow-up | Baseline, 3 months, 6 months
  Health-related quality of life will be measured using validated WHO-BREF Quality of life questionnaire.
Changes from baseline body mass index (BMI) at post intervention and 3 months follow-up. | Baseline, 3 months, 6 months
  Body weight (kilograms) and height (meters) will be combined and expressed as BMI (kg/m^2).
Changes from baseline body fat percentage at post intervention and 3 months follow-up | Baseline, 3 months, 6 months
  Body fat percentage will be estimated using a body composition analyser (In-Body, Korea).

OTHER OUTCOMES:
Intervention Adherence | 3 months
  Measure of Intervention adherence will based on participant attendance which is done by collecting given peer support posters, at the post-intervention level.
Socio-demographic characteristics | Baseline
  A brief questionnaire will be administered at the baseline to gather information on sociodemographic characteristic of participants including their age, gender, ethnicity and income levels.
Intervention Acceptance | 3 months
  Measure of acceptance will be measured using a short questionnaire which contains a series of three point scales scoring at the post-intervention level.

CONTACTS AND LOCATIONS:
Overall Officials: Amutha Ramadas, PhD, Principal Investigator — Monash University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03417128/Prot_SAP_000.pdf